CLINICAL TRIAL: NCT05223933
Title: Randomized Cluster Trial to Measure the Effectiveness of Home Care in Hyperendemic Rural Areas in Madagascar
Brief Title: Proactive Community Case Management (Pro-CCM) in Rural Madagascar
Acronym: Pro-CCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur de Madagascar (Other)
Collaborators: Peace Corps (Other); National Malaria Control Programme, Madagascar (Other Government); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rila Ratovoson, Researcher, Institut Pasteur de Madagascar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017-01
Record Dates: First submitted 2022-01-10; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Malaria; Case Management
Keywords: Malaria; Rural area; Community health workers
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: The study was a two-arm cluster randomized community intervention trial, with 11 fokontany in the intervention arm implementing malaria pro-CCM and 11 in the control arm. In both arms, CHWs provided passive integrative community case management (iCCM) among children under five per usual standard of care, including diagnosis with RDT for febrile illness, treatment with artesunate-amodiaquine according to RDT results, along with diagnosis and management of acute respiratory infections and diarrhea, and referral to a higher level of care if indicated. Oral rehydration salts, antibiotics were distributed to CHWs in the intervention arm to reinforce the iCCM activities already implemented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention fokontany (Experimental)
  Interventions: Behavioral: Proactive community case management
- Control fokontany (No Intervention)

INTERVENTIONS:
Behavioral: Proactive community case management — CHWs in the intervention arm conducted door-to-door fever screening for all inhabitants of all consenting households in their catchment area every fortnight. All individuals with temperature ≥ 37.5°C or history of self-reported fever in the previous two weeks were tested with an RDT; positive individuals who were not pregnant and did not have signs of severe disease were treated with artesunate-amodiaquine according to treatment guidelines. Individuals identified as requiring a referral during Pro-CCM visits were assisted with transfer to the healthcare center, with transportation handled by the project staff.
  Arms: Intervention fokontany

SUMMARY:
The trial took place in a rural area hyper endemic for malaria, the hypothesis of which was that active detection and treatment of malaria in the population (all ages combined) in the event of a positive test could reduce the prevalence of malaria in the region. zoned. It was a two-armed, randomized, cluster-based community intervention trial:

* one arm with home treatment of malaria for the duration of the study for patients with a positive result in the rapid diagnostic test for malaria.
* a control arm with the usual malaria management procedures (ie consultation with community workers or the nearest health centers in the event of fever or suspected signs of malaria).

Before the start of monitoring, an initial survey (Baseline) was carried out in the "fokontany" (villages / cluster) included in the 2 arms, in order to determine the prevalence of malaria. Then, in the intervention arm, screening for malaria by RDT every 2 weeks in subjects with a suspected malaria case (fever or notion of fever in the 2 days preceding the visit) and treatment with Artesunate-amodiaquine (ACT) for patients with a positive RDT. At the end of the follow-up period, a final survey (Endline), based on the same questionnaires as during the Baseline, was carried out in the 2 villages of the 2 arms.

As a secondary objective, a study on anemia in women aged between 15 and 49 years was also carried out during the baseline and endline periods in order to compare the prevalence between the 2 periods

DETAILED DESCRIPTION:
This study aims to compare the prevalence of malaria in the rural community of Mananjary after the Malaria Home Care Program (PECADOM Plus).

The study will take place in fokontany rural communes of the district of Mananjary.

This district was chosen for the following reasons:

* High prevalence of malaria in this area (31% in subjects with fever and attending medical consultation in the CSB included in the sentinel IPM fever site)
* presence of Peace Corps Volunteers (PCV) in this district. Mananjary District is situated in southeastern Madagascar, located in the central part of the Vatovavy Fitovinany Region, in the province of Fianarantsoa. It is located at 21°13'52" South and 48°20'31" East. The district is composed of one urban commune and 28 rural communes. After obtaining the agreement of the ethics committee for the realization of the study, the coordinator or the assistant coordinator of the project will make courtesy visits to all administrative and health officials in the Vatovavy Fitovinany and Mananjary District (Regional Directorate, District Chief ...).A random draw of fokontany meeting the inclusion criteria will be carried out later, to identify the distribution of fokontany in the intervention arm and control arm in the project. In addition to the 22 fokontany required, a draw of 8 reserve fokontany will be made (4 for each arm).

A courtesy visit will be conducted in the fokontany raffled. The coordinator will check the number of inhabitants in these fokontany with the information gathered at the time of the preparation of the protocol (projection of the population according to the data of INSTAT, information from the Medical Inspector of Mananjary). If the fokontany will not be eligible, the reserve fokontany will replace them in the study.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria in community:

  * Fokontany in rural communes of Mananjary district (fokontany level of safety, accessibility by the study teams, and phone network availability was assessed).
  * Agreement of the chief of Fokontany for the participation of his fokontany in the study
  * Fokontany with at least 1,000 inhabitants
* Individual inclusion criteria:

  * Resident in the relevant areas during the study period and consenting to participate

Exclusion Criteria:

* Exclusion criteria in community:

  * Fokontany with a total population of less than 1000 inhabitants
  * Fokontany in an urban commune
  * Fokontany in an area whose access is risky and perilous
* Individual exclusion criteria:

None (Non-resident present at the time of passage were tested in the study if they have suggestive signs of malaria but they were considered as visitors)

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2018-12-29 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study was the change in the prevalence of malaria RDT positivity in the intervention versus control fokontany. | an average of 1 year
  Difference in differences (DiD) approach comparing baseline to endline is used to compare the prevalence of malaria RDT positivity in the 2 arms

SECONDARY OUTCOMES:
percent of households visited every two weeks | The event was assessed up to 30 weeks (15 biweekly visits).
  percent of households visited every two weeks out of the number of the households registered in initial census
percent of households gave consent | The event was assessed up to 30 weeks (15 biweekly visits).
  percent of households that were visited every two weeks and gave consent for the screening during each visit
Fever incidence | The event was assessed up to 30 weeks (15 biweekly visits).
  percent of fever cases out of all individuals screened during each visit
Malaria incidence | The event was assessed up to 30 weeks (15 biweekly visits).
  percent of persons with positive RDT and fever cases out of all individuals screened during each visit
fever cases with RDT performed | The event was assessed up to 30 weeks (15 biweekly visits).
  percent of fever cases with RDT performed
RDT-positive persons treated with an ACT | The event was assessed up to 30 weeks (15 biweekly visits).
  percent of RDT-positive persons treated with an ACT during each visit
The change in the prevalence of anemia in women aged between 15 and 49 years old in the intervention versus control fokontany | an average of 1 year
  Difference in differences (DiD) approach comparing baseline to endline is used to compare the prevalence of anemia in the 2 arms

CONTACTS AND LOCATIONS:
Overall Officials: Rila Ratovoson, MD, Principal Investigator — Institut Pasteur de Madagascar; Milijaona Randrianarivelojosia, PhD, Study Director — Institut Pasteur de Madagascar
Locations (22):
- Madagascar (22):
  - Fokontany Andranomavo, Mananjary, : Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Ambakoana, Mananjary, Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Ambalamanasa, Mananjary, Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Ambalaromba, Mananjary, Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Ambinany Namorona, Mananjary, Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Amboditandroho, Mananjary, Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Ambohimiarina II, Mananjary, Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Ambohinihaonana, Mananjary, Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Ambolotara, Mananjary, Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Andranomiteka, Mananjary, Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Anilavinany, Mananjary, Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Ankazotokana, Mananjary, Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Anosimparihy, Mananjary, Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Kianjavato, Mananjary, Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Mahavoky Sud, Mananjary, Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Manotro, Mananjary, Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Maroamboka, Mananjary, Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Sahafotahina, Mananjary, Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Sandravakoka, Mananjary, Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Tanambao Sud, Mananjary, Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Tanambaobe, Mananjary, Fianarantsoa, Vatovavy Fitovinany
  - Fokontany Tsarahafatra, Mananjary, Fianarantsoa, Vatovavy Fitovinany

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Some summary data are available from December 2021; and some data at the time of publication (2022)
Access Criteria: IPD and any additional supporting information will be shared in supplementary files in publication and via Harvard Dataverse
URL: https://dataverse.harvard.edu/dataset.xhtml?persistentId=doi:10.7910/DVN/IIDE2B

REFERENCES:
- [Derived] Ratovoson R, Garchitorena A, Kassie D, Ravelonarivo JA, Andrianaranjaka V, Razanatsiorimalala S, Razafimandimby A, Rakotomanana F, Ohlstein L, Mangahasimbola R, Randrianirisoa SAN, Razafindrakoto J, Dentinger CM, Williamson J, Kapesa L, Piola P, Randrianarivelojosia M, Thwing J, Steinhardt LC, Baril L. Proactive community case management decreased malaria prevalence in rural Madagascar: results from a cluster randomized trial. BMC Med. 2022 Oct 4;20(1):322. doi: 10.1186/s12916-022-02530-x. PMID 36192774